CLINICAL TRIAL: NCT05916807
Title: Comparative Effects Of Stabilization Exercises And Posture Training On Pain Function And Range Of Motion In Breast Feeding Females Suffering From Scapular Dyskinesia
Brief Title: Effects of Stabilization Exercises and Posture Training on Breast Feeding Females Suffering From Scapular Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ashley Nudrat
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Scapular Dyskinesis
Keywords: Breast feeding; Pain; Range of motion; Scapular dyskinesis
MeSH Terms: conditions — Breast Feeding; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization Exercises (Experimental): Twenty-six (26) patients will be treated with stabilization exercises in breast feeding females suffering from scapular dyskinesia.
  Interventions: Other: Stabilization Exercises
- Posture Training (Experimental): Twenty-six (26) patients will be treated with posture training of breast-feeding females suffering from scapular dyskinesia.
  Interventions: Other: Posture Training

INTERVENTIONS:
Other: Stabilization Exercises — It consists of 26 patients who will receive stabilization exercises which will be divided in three components in lying posture, sitting, standing, rolling and kneeling positions to treat posterior, inferior muscles of scapula for 35-45 min for 3 days a week for 4 weeks.
  Arms: Stabilization Exercises
Other: Posture Training — It consists of 26 patients who will receive postural training and breast-feeding patterns for the mother and child for 35-45 min in 3 days a week for 4 weeks.
  Arms: Posture Training

SUMMARY:
A randomized clinical trial study will be conducted through a non-probability convenience sampling technique. Study will be conducted at Jinnah Hospital, Lahore. Sample size will be collected through open epi tool. The total sample size of 52 is calculated. Two treatment groups will be taken for conducting the research. Group A with twenty-six (26) patients will be treated with stabilization exercises and Group B with twenty-six (26) patients whom will be treated with posture training. Difference between pre-treatment and post-treatment readings will be calculated using Paired sample t-test for parametric data. For nonparametric data Wilcoxon signed rank test will be used. This is a non-parametric test that compares paired groups. Generalized physiotherapy rehabilitation protocol will be implemented in Group A for scapular stabilization by demonstrating scapular retraction (Shoulder Blade Squeezes), External Rotation, Shoulder Diagonals, Horizontal Rows, Shoulder Extension, Angel Wings, Active: Push with a plus, Physio ball Scapular Exercises, Platform Walks. In Group B, postural training different nursing positions will be guided as crossover hold, laid-back position, on the pillow position, cradle, football hold, side-lying position. The intervention will be provided in twelve sessions over a 4-week intervention period (three sessions per week) each session of 30 to 50 minutes accompanied by an individual daily at-home exercise program. The participants were advised not to use other forms of treatment during the trial (pharmacologic or non-pharmacologic treatment). NPRS will be used to measure the pain intensity and functional limitation will be assessed using the UEFI, goniometer to check the range limitation. Total study duration will be ten months after the approval of synopsis. Data will be analysed by using SPSS 26.

DETAILED DESCRIPTION:
Scapular dyskinesis is a change or deviation in the normal resting or active position of the scapula during shoulder movement due to the repetitive use of the shoulder, most people's scapula moves abnormally. Scapular winging is a clinical observation in which any part of the scapular departs excessively from the thorax soon after movement begins causing hinderance in performing movements like Elevation/depression, Protraction/retraction, Internal/external rotation, Superior/inferior rotation, Anterior/posterior tilt. Scapular dyskinesia can be caused by one of three factors, Shoulder-related, Neck-related, Posture-related.

The significance of this study is to lessen the musculoskeletal disorders causing scapular dyskinesia through provision of the stabilization, stretching exercises and posture training, improving function and range of motion in breast feeding females.

ELIGIBILITY:
Inclusion Criteria:

* Positive Scapular Dyskinesis Test
* Age 25-40 Years
* Breast feeding females from last 6 months
* Primigravida females

Exclusion Criteria:

* Cesarean section females
* Neck or shoulder pain due to any other comorbidity e.g. Previous history of trauma or fracture
* Any spinal deformity like scoliosis or kyphosis
* Disc prolapse facet joint stenosis

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | 4th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a one dimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases. Validity 0.86 to 0.95
UPPER EXTREMITY FUNCTIONAL INDEX | 4th week
  The Upper Extremity Functional Index is a patient reported outcome measure used to assess the functional impairment in individuals with musculoskeletal upper limb dysfunction.
RANGE OF MOTION | 4th Week
  A goniometer is an instrument that measures the available range of motion at a joint. The art and science of measuring the joint ranges in each plane of the joint are called goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panagiotopoulos AC, Crowther IM. Scapular Dyskinesia, the forgotten culprit of shoulder pain and how to rehabilitate. SICOT J. 2019;5:29. doi: 10.1051/sicotj/2019029. Epub 2019 Aug 20. PMID 31430250
- [Background] de Carvalho SC, Castro ADAE, Rodrigues JC, Cerqueira WS, Santos DDCB, Rosemberg LA. Snapping scapula syndrome: pictorial essay. Radiol Bras. 2019 Jul-Aug;52(4):262-267. doi: 10.1590/0100-3984.2017.0226. PMID 31435089
- [Background] Ezeukwu OA, Ojukwu CP, Okemuo AJ, Anih CF, Ikele IT, Chukwu SC. Biomechanical analysis of the three recommended breastfeeding positions. Work. 2020;66(1):183-191. doi: 10.3233/WOR-203162. PMID 32417825